

#### **FINAL**

November 16, 2022

# **Letter of Amendment 2**

**Protocol** 

Version 1.0

# **HVTN 139**

A phase 1 clinical trial to evaluate the safety and immunogenicity of HIV-1 vaccines based on chimpanzee serotypes of adenovirus expressing clade C gp140 and a CH505TF gp120 protein boost in healthy, HIV- uninfected adult participants

**DAIDS-ES ID 12052** 

A non-IND study

# HIV Vaccine Trials Network (HVTN) Clinical Research Site (CRS) filing instructions

The following information impacts the HVTN 139 study and must be forwarded to your Institutional Review Board (IRB)/Ethics Committee (EC) and any other applicable Regulatory Entity (RE) as soon as possible for their information and review. Their approval is required before implementation.

Upon receiving final IRB/EC and any other RE approval(s) for this Letter of Amendment (LOA), CRSs must implement the LOA immediately.

Upon receiving final IRB/EC and any other applicable RE approval(s), CRSs are required to submit LOA registration documents to the DAIDS Protocol Registration Office (PRO) at the Regulatory Support Center (RSC). CRSs will receive an LOA Registration Notification once the DAIDS PRO verifies that all the required LOA registration documents have been received and are complete. A Registration Notification from the DAIDS PRO is not required prior to implementing the LOA. A copy of the LOA Registration Notification, along with this LOA and any IRB/EC and RE correspondence, should be retained in the CRS's regulatory files.

For additional information on the registration process and specific documents required for LOA registration, refer to the current version of the DAIDS Protocol Registration Manual.

The following information does not affect the sample informed consent. The CRS's IRB/EC is responsible for determining the process of informing study participants of the contents of this LOA.

# List of changes

| Item 1 | Revised in Section 5, <i>Objectives and endpoints</i> : secondary objective 4 moved to exploratory objective 5 | 2 |
|---|---|---|
| Item 2 | Updated in Section 1.1, <i>Protocol Team</i> : Team membership, contact information, and roles | 3 |

The changes described herein will be incorporated in the next version of Protocol HVTN 139 if it undergoes full protocol amendment at a later time. Added text is shown in **bold underline** and deleted text is shown with **strikethrough**.

# Item 1 Revised in Section 5, *Objectives and endpoints*: secondary objective 4 moved to exploratory objective 5

The secondary objective 4 has been moved to exploratory objective 5 since the assay data is not being used for clinical management of the participant. It will be used for research purposes only. Results may be used to identify pre-existing immunity that may interfere with other key immunology assessments.

### Tracked revised text in section 5.2: Secondary objectives and endpoints

Secondary objective 4:

To evaluate vector-specific antibodies both before and after vaccination.

Secondary endpoint 4:

Magnitude of serum antibody neutralization of AdC6 and AdC7 vectors as assessed by adenovirus neutralization assay at baseline (Parts A and B), 4 weeks after the first vaccination (Parts A and B), and 4 weeks after the second vaccination (Part B)

## Tracked revised text in section 5.3: Exploratory objectives

#### Exploratory objective 5:

To assess the magnitude of serum antibody neutralization of AdC6 and AdC7 vector both before and after vaccination.

#### Item 2 Updated in Section 1.1, Protocol Team: Team membership, contact information, and roles

The Protocol Team list has been updated in Section 1.1, Protocol Team. Tracked revised text is shown below. Updated protocol team list is appended.

#### Tracked revised text under *Protocol leadership:*

Protocol Team leader

William Hahn Manuel

Villaran

HVTN LOC, Fred Hutch <del>206-667-3431</del> **206-667-675**7 whahn@fredhutch.org mvillar2@fredhutch.org

### Tracked revised text under other contributors to the original protocol:

LOC medical monitor

William Hahn Manuel

Villaran

HVTN LOC, Fred Hutch <del>206-667-3431</del> **206-667-6757** whahn@fredhutch.org

mvillar2@fredhutch.org

Clinical trials manager

Julie Hunt Taylor Jones-Bradford

**Nelisiwe Xaba** Michelle Nebergall HVTN LOC, Fred Hutch

Clinical data manager

Andrea Repetto, Bhavesha O'Byrne

HVTN SDMC, Fred Hutch

Statistical research Hua Zheng Xue Han

associate HVTN SDMC, Fred Hutch

Laboratory Center Representative Lisa Sanders Jen Hanke HVTN Laboratory Center,

Fred Hutch

Associate Director of

Regulatory affairs

Megan Brandon

HVTN LOC, Fred Hutch

Protocol development managers

Rufi Dalvi Kajari Mondal

Daciana Margineantu HVTN LOC, Fred Hutch Project coordinator

**Anders McConachie** Haven Wilvich

HVTN LOC, Fred Hutch

#### 1.1 **Protocol Team** Protocol leadership

Chair Ameena Goga Statistician Youyi Fong

HIV Prevention Research Unit, HVTN SDMC, Fred Hutch

South African Medical Research 206-667-1093 Council yfong@fredhutch.org

Ameena.Goga@mrc.ac.za

+2712 339 8524 +2782 302 3168

Steven Innes DAIDS Medical Edith Swann Co-chair

> Emavundleni Research Centre DAIDS, NIAID officer +27 21 650 5851 240-627-3035

+27 74 764 5253 301-332-6435-BB Steven.Innes@hiv-research.org.za swanne@niaid.nih.gov

Protocol Team leader Manuel Villaran Stephen De Rosa Laboratory lead

HVTN LOC, Fred Hutch **HVTN Laboratory Center** 

206-667-6757 206-667-1681 mvillar2@fredhutch.org sderosa@fredhutch.org

#### Other contributors to the original protocol

Michael Pensiero LOC medical monitor DAIDS Product Lead Manuel Villaran DAIDS, NIAID

HVTN LOC, Fred Hutch 301-435-3749 206-667-6757

mpensiero@niaid.nih.gov mvillar2@fredhutch.org

Oladapo Alli Study product Hildegund Ertl DAIDS protocol DAIDS, NIAID developer Wistar Institute Vaccine and pharmacist

240-627-3593 representatives Immunotherapy Center

> Emmanuel (Chip) Walter April Randhawa SDMC Associate

Duke Human Vaccine Institute HVTN SDMC, Fred Hutch director of lab science

Zachary Sagawa Infectious Disease Research

Institute

Research Council

Taylor Jones-Bradford Laboratory Center Jen Hanke Clinical trials manager

HVTN Laboratory Center, Representative Michelle Nebergall Fred Hutch HVTN LOC, Fred Hutch

Maija Anderson Associate Director of Clinical safety specialist Megan Brandon

Regulatory affairs HVTN LOC, Fred Hutch HVTN LOC, Fred Hutch

Community engagement Regional Medical Liaison Azwi Takalani Baepanye Kagisho

unit representative HVTN LOC, Fred Hutch HVTN LOC, Fred Hutch

Clinic coordinator **Brodie Daniels** Community Mduduzi Ngubane

educator/recruiter Isipingo South African Medical Isipingo South African Medical

Research Council Research Council

Community Advisory Sphelelo Mqadi Clinical data manager Andrea Repetto,

Isipingo South African Medical Board (CAB) member HVTN SDMC, Fred Hutch

> Rufi Dalvi Statistical research Xue Han

Kajari Mondal HVTN SDMC, Fred Hutch managers associate

HVTN LOC, Fred Hutch

Anders McConachie Project coordinator

HVTN LOC, Fred Hutch

Nelisiwe Xaba

Protocol development

# **Protocol modification history**

Protocol modifications are made to HVTN protocols via clarification memos, letters of amendment, or full protocol amendments. HVTN protocols are modified and distributed according to the standard HVTN procedures as described in the HVTN Manual of Operations (MOP).

The version history of, and modifications to, Protocol HVTN 139 are described below.

#### Date: November 16, 2022

Protocol version: Version 1.0

Protocol modification: Letter of Amendment 2

- Item 1 Revised in Section 5, *Objectives and endpoints*: secondary objective 4 moved to exploratory objective 5
- Item 2 Updated in Section 1.1, *Protocol Team*: Team membership, contact information, and roles

# Date: May 19, 2022

Protocol version: Version 1.0

Protocol modification: Clarification Memo 2

Item 1 Updated in Appendix H, Laboratory procedures Part B; Appendix J, Procedures at HVTN CRS for Part B; and Appendix L, HVTN 139 Visit Windows for Part B: visit numbers for Part B

#### Date: March 07, 2022

Protocol version: Version 1.0

Protocol modification: Clarification Memo 1

Item 1 Updated in Section 8.3.1, AdC6-HIVgp140; Section 8.3.2, AdC7-HIVgp140; and 8.3.4, Placebo for AdC6-HIVgp140 and AdC7-HIVgp140: label of study products

#### Date: June 15, 2021

Protocol version: Version 1.0

Protocol modification: Letter of Amendment 1

- Item 1 Revised in Section 4.10.1, Clinical studies of Chimpanzee Ad vectors targeting diverse pathogens, Section 4.11, Potential risks of study products and administration, Appendices A and B, Sample Informed Consent Form for Part A and Part B (section 4), and Appendix N, Adverse events of special interest: risks of AdC6 and AdC7 study products
- Item 2 Revised in *Appendix A, Sample Informed Consent Form for Part A,* Sections 4 and 17: study product developer information

- Item 3 Revised in Appendix B, Sample Informed Consent Form for Part B, Section 4: study product developer information
- Item 4 Revised Section 1.1, *Protocol Team, Protocol Team Leadership:* Co-Chair and member contact information
- Item 5 Clarified in Section 9, *Clinic Procedures:* procedures for data entry into the study database and reference to the HVTN HIV testing algorithm
- Item 6 Clarified in Section 12, Protocol conduct: protocol monitoring
- Item 7 Updated Section 14, *Document references (other than literature citations):* the URL for requirements for source documentation

# Date: February 23, 2021

Protocol version: Version 1.0 Protocol modification: N/A

Original protocol

# Protocol signature page

A phase 1 clinical trial to evaluate the safety and immunogenicity of HIV-1 vaccines based on chimpanzee serotypes of adenovirus expressing clade C gp140 and a CH505TF gp120 protein boost in healthy, HIV- uninfected adult participants.

I will conduct the study in accordance with the provisions of this protocol and all applicable protocol-related documents. I agree to conduct this study in compliance with United States (US) Health and Human Service regulations (45 CFR 46); applicable US Food and Drug Administration regulations; standards of the International Conference on Harmonization Guideline for Good Clinical Practice (E6); Institutional Review Board/Ethics Committee determinations; all applicable in-country, state, and local laws and regulations; and other applicable requirements (eg, US National Institutes of Health, Division of AIDS) and institutional policies.

Investigator of Record Name (print)

Investigator of Record Signature

Date

DAIDS Protocol Number: HVTN 139

DAIDS Protocol Version: Version 1.0

Protocol Date: February 23, 2021